CLINICAL TRIAL: NCT06907238
Title: The Value of Novel Thrombus Markers in the Diagnosis and Treatment of Acute Pulmonary Embolism
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 3308872
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Acute Pulmonary Embolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- APE group
- non APE group

SUMMARY:
In response to the high mortality rate of patients with acute pulmonary embolism (APE) and the fact that only a small proportion of deceased patients can receive correct diagnosis, this study will use a sensitive, non-invasive, and feasible new thrombus molecular marker (TAT/PIC/TM/t-PAIC) to detect and evaluate the activation of the coagulation and fibrinolysis systems and endothelial system damage in patients, in order to monitor the early diagnosis and treatment of APE, reduce mortality, and improve patient quality of life. Therefore, this study intends to include 200 newly diagnosed APE patients to evaluate the sensitivity and specificity of the single and combined application of novel thrombus molecular markers for APE diagnosis; Detect the biomarker results of patients at different time points before and after treatment, and evaluate their value in APE treatment monitoring; Track and follow up on patients after discharge to explore the prognostic value of biomarkers for APE.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients diagnosed with APE for the first time through CTPA in clinical practice and who have not received anticoagulant therapy in the past month; 2.Age ≥ 18 years old.

Exclusion Criteria:

* 1. Complicated with other thrombotic diseases, complicated with important organ damage such as heart, liver, kidney, and previous history of pulmonary embolism; 2. Malignant tumors; 3. Renal dialysis patients; 4. Antiphospholipid syndrome; 5. Immune system diseases; 6. Hematological diseases; 7. DIC caused by severe infection; 8. Patients judged by clinicians to be unfit for clinical practice.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients in APE group and 200 patients in non APE group each
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-10-14 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
New thrombusmarkers (TAT/PIC/TM/t-PAIC) | Data of patients on the first, the fourth day, seventh and tenth days after admission for diagnosis. If the duration of hospitalization is ≤ 7 days, data will be collected only three times

SECONDARY OUTCOMES:
Conventional coagulation indicators, PT、APTT、FIB、D-Dimer and FDP | Data of patients on the first, the fourth day, seventh and tenth days after admission for diagnosis. If the duration of hospitalization is ≤ 7 days, data will be collected only three times

IPD SHARING:
Plan to Share IPD: No